CLINICAL TRIAL: NCT07328074
Title: Prospective Cohort Study of Electrocautery Resection Combined With Hyperthermic Intrathoracic Chemotherapy for Thymic Epithelial Tumors With Pleural Metastasis
Brief Title: Electrocautery Resection Combined With HITHOC for Thymic Epithelial Tumors With Pleural Metastasis
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Jiang Fan, Professor, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Other Study IDs: 20250519101831997
Record Dates: First submitted 2025-12-28; First posted 2026-01-08 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-12

CONDITIONS: Thymic Epithelial Tumor; Thymoma; Thymic Carcinoma; Pleural Metastasis; Pleural Recurrence
Keywords: Hyperthermic Intrathoracic Chemotherapy; HITHOC; Electrocautery; Cisplatin; Doxorubicin
MeSH Terms: conditions — Thymic epithelial tumor; Thymoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Electrocautery Resection + HITHOC: Patients with thymic epithelial tumors with pleural metastasis or recurrence who undergo extended thymectomy with electrocautery resection of pleural metastases followed by two cycles of hyperthermic intrathoracic chemotherapy (HITHOC) with cisplatin and doxorubicin.
  Interventions: Procedure: Patients with thymic epithelial tumors with pleural metastasis or recurrence who undergo extended thymectomy with electrocautery resection of pleural metastases followed by two cycles of hyperthermic; Procedure: Hyperthermic Intrathoracic Chemotherapy (HITHOC)

INTERVENTIONS:
Procedure: Patients with thymic epithelial tumors with pleural metastasis or recurrence who undergo extended thymectomy with electrocautery resection of pleural metastases followed by two cycles of hyperthermic — Extended thymectomy with electrocautery ablation and resection of pleural metastases. Larger lesions (>1cm) are thoroughly ablated with electrocautery followed by complete resection. Smaller lesions (≤1cm) that are difficult to resect are thoroughly ablated with electrocautery.
Procedure: Hyperthermic Intrathoracic Chemotherapy (HITHOC) — Two cycles of hyperthermic intrathoracic chemotherapy performed 2-4 days apart using BR-TRG-I device. Chemotherapy solution containing cisplatin (50 mg/m²) and doxorubicin (25 mg/m²) is circulated at 400 mL/min with inflow temperature maintained at 42-43°C for 60 minutes per cycle.

SUMMARY:
The goal of this observational study is to explore the effectiveness of electrocautery resection combined with hyperthermic intrathoracic chemotherapy (HITHOC) in patients with thymic epithelial tumors with pleural metastasis or recurrence. The study aims to:

* Evaluate whether this combined treatment improves event-free survival in patients with pleural metastasis from thymic epithelial tumors
* Assess the rates of grade ≥3 treatment-related adverse events
* Examine how this treatment affects patients' quality of life

Participants will:

* Undergo extended thymectomy with electrocautery resection of pleural metastases
* Receive two cycles of hyperthermic intrathoracic chemotherapy with cisplatin and doxorubicin at 42-43°C, 2-4 days apart
* Complete quality of life questionnaires (EQ-5D) at baseline and regular intervals
* Have regular follow-up visits with imaging and clinical assessments for up to 36 months to monitor for disease recurrence or progression

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed thymic epithelial tumor (TET)
* Imaging evidence of thymic epithelial tumor with pleural dissemination or recurrence, deemed suitable for HITHOC by multidisciplinary thoracic team
* Age ≥16 years and ≤80 years
* American Society of Anesthesiologists (ASA) physical status classification I-II
* Normal major organ function
* No history of other malignancies
* Prior chemotherapy completed >4 weeks, radiotherapy >6 weeks, immunotherapy >6 weeks before enrollment
* No allergy to cisplatin or doxorubicin
* Able to understand the study content and provide informed consent

Exclusion Criteria:

* Evidence of extrathoracic metastasis on imaging or pathological examination
* Myasthenia gravis in unstable phase or acute exacerbation
* Severe systemic comorbidities, such as active infection, poorly controlled diabetes, coagulopathy, bleeding tendency, or ongoing thrombolytic/anticoagulation therapy
* Positive serum pregnancy test or lactation (females)
* History of organ transplantation (including autologous bone marrow transplantation and peripheral blood stem cell transplantation)
* History of peripheral nervous system disease, significant psychiatric disorder, or central nervous system disease
* Currently participating in other clinical trials

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adults aged 16-80 years with pathologically confirmed thymic epithelial tumors (thymoma or thymic carcinoma) with pleural dissemination or recurrence, suitable for electrocautery resection and hyperthermic intrathoracic chemotherapy as determined by multidisciplinary team.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2031-02 (Estimated); Study Completion 2031-02 (Estimated)

PRIMARY OUTCOMES:
Event-Free Survival (EFS) | From treatment initiation to first event (local recurrence, distant metastasis, or death), assessed up to 36 months
  Time from treatment start to first occurrence of local recurrence, distant metastasis, or death from any cause. Events are assessed through regular imaging and clinical follow-up.

SECONDARY OUTCOMES:
Incidence of Grade ≥3 Treatment-Related Adverse Events | From treatment initiation through 30 days post-treatment
  Rate of grade ≥3 adverse events according to Clavien-Dindo classification related to surgery or chemotherapy. This includes surgical complications and chemotherapy-related toxicities.
Overall Survival (OS) | From enrollment to death from any cause, assessed up to 36 months
  Time from disease grouping to death from any cause.
Quality of Life Assessed by EQ-5D | Baseline, post-treatment, and at 3, 6, 12, 24, and 36 months
  Quality of life assessed using the EuroQol 5 Dimensions (EQ-5D) questionnaire. The EQ-5D visual analog scale ranges from 0 (worst imaginable health state) to 100 (best imaginable health state). Higher scores indicate better quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai General Hospital, Department of Thoracic Surgery, Shanghai, Shanghai Municipality, China